CLINICAL TRIAL: NCT02916186
Title: Evaluation of Subepithelial Connective Tissue Graft Versus Acellular Dermal Matrix With Tunnel Technique in Treatment of Multiple Gingival Recessions (Randomized Clinical Trial, Parallel Design)
Brief Title: Evaluation of Subepithelial Connective Tissue Graft Versus Acellular Dermal Matrix With Tunnel Technique in Treatment of Multiple Gingival Recessions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatema Mohammed Ali Elmahdi, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-197
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tunnel technique with acellular dermal matrix (Experimental): the tunnel technique involves separation of the gingiva, then acellular dermal matrix interposed between the flap and the root surface.
  Interventions: Biological: Acellular Dermal Matrix; Procedure: Tunnel technique with the subepithelial connective tissue graft
- subepithelial connective tissue graft (Active Comparator): Tunnel is prepared and sub-epithelial connective tissue graft is harvested from the palate and placed under the flap.
  Interventions: Biological: Acellular Dermal Matrix; Procedure: Tunnel technique with the subepithelial connective tissue graft

INTERVENTIONS:
Biological: Acellular Dermal Matrix — Puros Dermis is a collagenous membrane derived from solvent preserved,human dermis, works as biological scaffold for the new formation of vasculated connective tissue.
  Other Names: Puros Dermis Allograft Tissue Matrix
Procedure: Tunnel technique with the subepithelial connective tissue graft — Tunnel prepared with the placement of subepithelial connective tissue graft harvested from the palate
  Other Names: autogenous connective tissue graft

SUMMARY:
The goal of the present study is to compare the amount of root coverage resulting from subepithelial connective tissue graft and acellular dermal matrix associated with tunnel technique among patients suffering from multiple gingival recession.

DETAILED DESCRIPTION:
Acellular dermal matrix with Tunnel technique will offers great advantages for patients with multiple gingival recession as regards decrease surgical time, Post-Operative pain and root coverage, clinical attachment level, width of Keratinized gingiva, gingival biotype compared to subepithelial connective tissue graft with Tunnel technique.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with facial multiple gingival recession defects classified as either class I or II defects according to Miller's classification (Miller 1985).
* Subjects aged between 18 - 60 years old.
* Patients should be free from any systemic disease that may affect normal healing of tissue, and predictable outcome.
* Patients with good oral hygiene.

Exclusion Criteria:

* Current and former smokers.
* Pregnant females.
* Subjects received any periodontal therapy for minimum of 6 months prior to the study.
* Subjects taking drugs known to interfere with wound healing.
* Subjects with unacceptable oral hygiene with plaque index >2.
* Teeth with non-carious cervical lesions (NCCL), cervical caries and malalignment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
patient Satisfaction . | 1 year
  measured by VAS scale

SECONDARY OUTCOMES:
root coverage | 1 year
  measured by periodontal probe
Clinical Attachment Level | 1 year
  measured by periodontal probe
Width of Keratinized Tissue | 1 year
  measured by periodontal probe
Gingival Bio-type | 1 year
  measured by endodontics file

IPD SHARING:
Plan to Share IPD: Undecided